CLINICAL TRIAL: NCT07187115
Title: A Global Randomized Trial Comparing Pulsed Field Ablation of Pulmonary Veins Plus Extra-PV Sources Utilizing Electrographic Flow Mapping Versus Pulmonary Veins Plus Posterior Wall in Persistent Atrial Fibrillation Patients.
Brief Title: A Global Study Comparing Pulsed Field Ablation With Electrographic Flow Mapping Versus Posterior Wall Ablation for Persistent Atrial Fibrillation
Acronym: OPTIMIZE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF334
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Persistant Atrial Fibrillation
Keywords: FARAPULSE; FARAPOINT; OptiMap
MeSH Terms: conditions — Atrial Fibrillation | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: plus non-randomized cohorts (Attempt, Roll-in)
Masking Description: The investigators and staffs will be blinded to the EGF maps in Control Arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control Arm (Active Comparator): PVI + PWA: The Control Arm, consisting of subjects undergoing PVI + PWA. PWA will be performed adjunctive to PVI per protocol Section 10.8.10. Following confirmation of PWA, EGF mapping will be performed in the LA and RA, while Investigators, lab/nursing staff, and research personnel are blinded to the EGF maps.
  Interventions: Device: OptiMap System (non-ablative); Device: FARAPULSE Pulsed Field Ablation (PFA) System and Opal HDx Mapping System
- Treatment Arm (Experimental): PVI + EGF source(s) ablation: The Treatment Arm, consisting of subjects undergoing PVI + EGF source(s) ablation. Adjunctive to PVI, the EGF-identified active sources above threshold will be ablated per protocol Section 10.8.11. If following PVI, a narrow channel that is approximately ≤ 1 cm is identified in the LAPW, ablation may be performed using the FARAPOINT Catheter.
  Interventions: Device: FARAPOINT Pulsed Field Ablation System; Device: OptiMap System (non-ablative); Device: FARAPULSE Pulsed Field Ablation (PFA) System and Opal HDx Mapping System

INTERVENTIONS:
Device: FARAPOINT Pulsed Field Ablation System — A component of the FARAPULSE Pulsed Field Ablation (PFA) System and is a multi-electrode bidirectional, deflectable percutaneous catheter, an adjunctive catheter designed to create focal-type lesions for the creation of an ablation line between the inferior vena cava and the tricuspid valve.
  Arms: Treatment Arm
Device: OptiMap System (non-ablative) — An electrophysiology mapping system that uses a proprietary algorithm to analyze electrogram signals.
  Other Names: Ablamap System
Device: FARAPULSE Pulsed Field Ablation (PFA) System and Opal HDx Mapping System — All subjects will undergo electroanatomical mapping of the entire left atrium with the FARAWAVE NAV Catheter and Opal HDx Mapping System, followed by PFA PVI with the FARAWAVE NAV PFA Catheter, per the instructions of use.

SUMMARY:
The purpose of this study is to establish the safety of the pulsed field ablation (PFA) therapy of Pulmonary Veins and Electrographic Flow (EGF) identified extra-PV sources of atrial fibrillation (PVI + EGF ablation of sources) and to demonstrate its non-inferiority in effectiveness compared to PFA of Pulmonary Veins and LA Posterior Wall (PVI+ PWA) in the treatment of de novo symptomatic drug-refractory persistent atrial fibrillation (PersAF).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age, or older if required by local law
2. Have symptomatic drug-refractory1, persistent AF2, confirmed by both:

   * Documentation, such as physician note, of persistent continuous AF for > 7 days and ≤ 365 days and the arrhythmia symptoms
   * Documentation, within 180 days of enrollment date of either:

     * A 24-hour continuous ECG recording confirming continuous AF or
     * Two (2) ECGs (from any regulatory cleared rhythm monitoring device) showing continuous AF taken at least 7 days apart
3. Willing and capable of providing informed consent
4. Willing and capable of participating in all follow-up assessments and testing associated with this clinical investigation at an approved clinical investigational center
5. Willing to receive LUX-Dx™ insertable cardiac monitor (ICM) during the study or already has a LUX-Dx™ ICM that was inserted ≤ 6 months (i.e., within 180 days) of consent, and willing to comply to the LUX-Dx Latitude Clarity transmission instructions

Exclusion Criteria:

1. Any of the following atrial conditions:

   1. Left atrial anteroposterior diameter ≥ 5.5 cm, or if1 LA diameter not available, non-indexed volume >100 ml (physician note or imaging)
   2. Any prior left atrial ablation
   3. Any prior atrial surgery
   4. Current atrial myxoma
   5. Current left atrial thrombus
   6. Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
2. Any of the following cardiovascular conditions:

   1. History of sustained ventricular tachycardia or any ventricular fibrillation
   2. Severe right ventricular dysfunction with documented echocardiography and/or hemodynamic data, per Investigator's discretion
   3. AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
   4. Cardiac devices and implants:

      * Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices
      * Implantable loop recorder, other than LUX-Dx
      * Interatrial baffle, patent foramen ovale or atrial septal defect closure device or patch
      * Any left atrial appendage closure or occlusion device
   5. Presence of any of the following valvular conditions:

      * Any prosthetic heart valve, stenotic valves, ring or repair
      * Moderate to severe mitral valve stenosis
      * More than moderate mitral regurgitation
   6. Hypertrophic or amyloid cardiomyopathy
   7. Any IVC filter, known inability to obtain vascular access or other contraindication to femoral access
   8. Awaiting cardiac transplantation or other planned cardiac surgery within the next 12 months
   9. Severe right ventricular dysfunction with documented echocardiography and/or hemodynamic data.
3. Any of the following conditions at Baseline:

   1. Heart failure associated with NYHA Class III or IV
   2. Most recent documented LVEF < 40% within the previous 12 months
   3. Body Mass Index (BMI) > 45.0
   4. Known coagulopathy or bleeding disorder
   5. Contraindication to, or unwillingness to use systemic anticoagulation, or acceptable alternatives, pre-, intra- and post-procedure to achieve adequate anticoagulation
   6. Women who are confirmed to be pregnant or lactating at the time of the ablation procedure
   7. Severe lung disease, severe pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
   8. Active malignancy (other than squamous cell carcinoma)
   9. Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
   10. Known active systemic infection
   11. Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour) as per the guidelines
   12. Predicted life expectancy less than one year per investigator medical judgement
   13. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility
   14. Required use of phosphodiesterase inhibitors within 24 hours of the ablation procedure
   15. Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two (2) BP measurements at baseline assessment not attributable to white coat syndrome per Investigator opinion
   16. CHA2DS2-VASc score ≥ 5
   17. Known allergic drug reaction to nitroglycerin (excluding hypotension)
   18. Unwillingness to receive, or unable to tolerate, a subcutaneous, chronically inserted LUX-Dx ICM device
4. Any of the following congenital conditions:

   1. Congenital heart disease with any clinically significant residual anatomic or conduction abnormality
   2. History of known congenital methemoglobinemia
   3. History of known G6PD deficiency
5. Any of the following conditions in the medical history:

   1. Solid organ or hematologic transplant, or currently being evaluated for a transplant
   2. Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis
   3. Any documented history of Prinzmetal Angina or severe non-revascularizable coronary disease
   4. Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
   5. Any other general health condition that, in the investigator's medical opinion, would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation.
6. Any of the following events less than or equal to 90 days of the consent date:

   1. Myocardial infarction (MI), unstable angina or coronary intervention
   2. Any cardiac surgery
   3. Heart failure hospitalization
   4. Pericarditis or symptomatic pericardial effusion
   5. Gastrointestinal bleeding
   6. Stroke, TIA, or intracranial bleeding
   7. Any active non-neurologic thrombus and/or thromboembolic event
   8. Carotid stenting or endarterectomy
   9. Uncontrolled diabetes mellitus or a recorded HbA1c > 8.0%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 60 Days
  The primary safety endpoint is the rate of ITT subjects in the PVI+EGF arm with one or more of the following serious device- or procedure-related Composite Adverse Events (CAEs) assessed through 60 days following the Index Procedure.
Primary Effectiveness Endpoint | 365 Days
  The primary effectiveness endpoint is the rate of ITT subjects with treatment success in the PVI+EGF arm vs. the PVI+PWA control arm through Day 365, aiming to demonstrate non-inferiority of PVI+EGF compared to the PVI+PWA control.

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint | 365 Days
  The secondary effectiveness endpoint is a test for superiority in Treatment Success between the Treatment Arm and the Control Arm. The test for superiority will only be conducted if the non-inferiority test for the PEE is passed and the result favors the Treatment Arm.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (29):
  - Grandview Medical Center, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Banner University Medical Center, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Alta Bates Summit Medical Center, Oakland, California
  - Stanford University Medical Center, Palo Alto, California
  - Pacific Heart Institute, Santa Monica, California
  - Piedmont Athens Regional, Athens, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Endeavor Hospital, Glenview, Illinois
  - Mercy Hospital Medical Center, West Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Good Samaritan - Suffern, Suffern, New York
  - Mission Hospital, Asheville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Sacred Heart Medical Center at Riverbend, Springfield, Oregon
  - Presbyterian University of Pennsylvania Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Hartcentrum Hasselt Jessa Ziekenhuis Campus Virga Jesse, Hasselt
- Centre Hôpital Universitaire Rouen, Hôpital Charles Nicolle, Rouen, France
- MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt, Germany
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC - University Medical Center Rotterdam, Rotterdam
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre